CLINICAL TRIAL: NCT05748730
Title: The Center for Enhancing Triage and Utilization for Depression and Emergent Suicidality (ETUDES) in Pediatric Primary Care-iCHART RCT
Brief Title: Clinical Trial for Integrated Care to Help At Risk Teen (iCHART) Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Children's Hospital of Philadelphia (Other); University of Oregon (Other); Columbia University (Other); Kaiser Permanente (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stephanie Stepp, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY22020069; P50MH115838 (NIH)
Record Dates: First submitted 2023-02-08; First posted 2023-03-01 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Suicide and Depression; Adolescent Behavior
MeSH Terms: conditions — Suicide; Depression; Adolescent Behavior | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This study uses an effectiveness-implementation hybrid type 1 randomized clinical trial (RCT) design.
  A qualitative, descriptive design will be used to analyze qualitative aims of this study.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be masked to the intervention condition at follow-up assessment time points.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iCHART (Experimental): iCHART is an intervention that includes 3 components previously studied in within the ETUDES Center including a:
  1. Safety Planning App for suicidal youth which enables a primary care provider to streamline the gold standard of care for those with current suicidality symptoms through an app (instead of a paper based version);
  2. Mental Health Screener questionnaire that gathers additional mental health symptoms, treatment preferences, and family's readiness for treatment engagement to help primary care provider make a personalized, tailored treatment plan a suicidal youth is more likely to adhere to;
  3. Text Messages which aims to provide texts for 2-3 weeks to motivate you to engage with the safety plan and recommended treatment following the patient visit.
  Participants will receive usual care at their pediatric primary care practice following screening including information, psychoeducation, and referral to a mental health treatment provider.
  Interventions: Behavioral: iCHART
- Treatment As Usual (TAU) (Active Comparator): Participants in this group will receive usual care from their primary care provider or mental health care provider which may include development of a paper safety plan.
  Interventions: Behavioral: Treatment As Usual

INTERVENTIONS:
Behavioral: iCHART — The Safety Planning App will guide primary care providers or mental health clinicians in the use of an emotion regulation and safety planning app (BRITE) to be loaded on the phone of depressed and suicidal adolescents in order to improve depression and reduce the likelihood of a suicide attempt.
  The Mental Health Screener is a decision support tool to guide the primary care provider to make a referral that reflects patient clinical needs and patient and parental treatment preferences and perceived barriers to treatment.
  The Text Messages is a personalized text messaging intervention for patients and parents that targets engagement with the safety plan to increase the likelihood that a depressed or suicidal patient will maintain or initiate recommended services.
  Participants will receive usual care at their pediatric primary care practice following screening including information, psychoeducation, and referral to a mental health treatment provider.
  Arms: iCHART
Behavioral: Treatment As Usual — Participants in this group will receive usual care from their primary care provider or mental health care provider which may include development of a paper safety plan.
  Arms: Treatment As Usual (TAU)

SUMMARY:
This protocol will test the effectiveness of an intervention, iCHART (integrated Care to Help At-Risk Teens) and facilitate recruitment for other studies in the larger ETUDES Center grant, which are focused on treatment development for target risk factors for suicidal behavior, specifically, sleep, anhedonia, and stress related to cybervictimization. This study will recruit 900 adolescents which will be enrolled in a randomized controlled trial to test iCHART and will be randomized to iCHART or treatment as usual (TAU). Based on previous work, the investigators hypothesize that iCHART, compared to TAU, will decrease suicidal-related events by 50%, and the effects will be mediated by increases in referrals, treatment engagement, and safety planning. The investigators will use implementation science methods to assess contextual factors (i.e., barriers and facilitators) and implementation outcomes specifically, acceptability, feasibility, appropriateness, and cost for our predictive algorithm and iCHART to inform future implementation efforts and promote health equity.

DETAILED DESCRIPTION:
iCHART is an intervention that includes 3 components previously studied in within the ETUDES Center including the:

1. Safety planning app for suicidal youth which enables a primary care provider to streamline the gold standard of care for those with current suicidality symptoms through an app (instead of a paper based version);
2. Mental Health Screener questionnaire that gathers additional mental health symptoms, treatment preferences, and family's readiness for treatment engagement to help primary care provider make a personalized, tailored treatment plan a suicidal youth is more likely to adhere to;
3. Text Messages which aims to provide texts for 2-3 weeks to motivate youth to engage with the safety plan and recommended treatment following the patient visit.

Aim 1. Test the effectiveness of iCHART in reducing suicide-related events at 6 months, the primary outcome, and examine mediators and moderators of treatment response. The investigators hypothesize: 1) iCHART will reduce suicide-related events and its effects will be mediated by increases in mental health referrals made by pediatric providers (any designated staff member, doctor, nurse on the treatment team); treatment engagement (i.e., follow through with mental health referrals), and safety planning (as evident by EHR reviews); 2) Individual-, family-, and neighborhood-level risk and protective factors will moderate response; and 3) Examine a predictive algorithm to examine heterogeneity of treatment response.

Aim 2. Examine barriers, facilitators, and implementation outcomes specifically, acceptability, feasibility, appropriateness, and cost for the predictive algorithm and iCHART to inform future implementation efforts and promote health equity. Barriers and facilitators that span multiple levels of context (e.g., aspects of clinic workflows, provider beliefs and knowledge) are expected to be uncovered. Further, incorporating the predictive algorithm and iCHART in pediatric primary care will be viewed as feasible, acceptable, and appropriate by youth, caregivers, and providers across different racial and ethnic groups.

ELIGIBILITY:
Inclusion Criteria:

* YOUTH

  * Youth will be age 12-18 and speak English.
  * Youth will have current depression or suicidal behavior. Suicidal behavior for iCHART (N=900) is defined as past suicidal thoughts in the past two weeks as indicated by PHQ-9M item #9 ≥ 1, and/or past month suicidal thoughts, and/or prior history of attempt as indicated by items on the PHQ-9M; and 300 who screen positive for depression (PHQ-9M ≥ "11")
  * 50% of the 300 youth with PHQ-9M ≥ "11" will also be positive for suicide risk as defined for iCHART.
* CAREGIVERS/PARENTS

  * Parents/caregivers of youth in the study must be at least 18 years old and their child must be willing to participate in the study. Caregivers/parents must be able to speak English. Parents are considered biological/adoptive parents or have court documentation that they can provide consent for research as a legal guardian of a youth. Only 1 parent/caregiver will be engaged in research, but in case 1 parent is unavailable, the other may be engaged (meaning it doesn't have to be the same parent participating in assessments/interviews throughout youth study participation).

Exclusion Criteria:

* YOUTH

  * Exclusion criteria include conditions that might impair their ability to effectively deploy ETUDES interventions, including:
  * current manic or psychotic episode, presence of a life-threatening medical condition requiring immediate treatment, intellectual or developmental disability precluding comprehension of study procedure. The latter will will be assessed by parental report of placement in self-contained Special Education classes, EHR review, and during the consent/assent and/or baseline to determine if the participant is not understanding research procedures.
  * Participants without access to a phone and/or tablet to interact with components of the intervention that require a phone will be excluded.
* CAREGIVERS/PARENTS

  * There are no specific exclusion criteria for caregivers and providers. However, as mentioned in the inclusion criteria, caregivers will be excluded if they are not the biological parent or court-appointed guardian of the youth being interviewed.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 900 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Depression Severity | Baseline
  Total scores from the Patient Health Questionnaire (PHQ-9-M) will be used to assess depression severity. Total Score Depression Severity: 0-4 No or Minimal depression; 5-9 Mild depression; 10-14 Moderate depression; 15-19 Moderately severe depression; 20-27 Severe depression.
Depression Severity | 1 Month Follow Up
  Total scores from the Patient Health Questionnaire (PHQ-9-M) will be used to assess depression severity. Total Score Depression Severity: 0-4 No or Minimal depression; 5-9 Mild depression; 10-14 Moderate depression; 15-19 Moderately severe depression; 20-27 Severe depression.
Depression Severity | 3 Month Follow Up
  Total scores from the Patient Health Questionnaire (PHQ-9-M) will be used to assess depression severity. Total Score Depression Severity: 0-4 No or Minimal depression; 5-9 Mild depression; 10-14 Moderate depression; 15-19 Moderately severe depression; 20-27 Severe depression.
Depression Severity | 6 Month Follow Up
  Total scores from the Patient Health Questionnaire (PHQ-9-M) will be used to assess depression severity. Total Score Depression Severity: 0-4 No or Minimal depression; 5-9 Mild depression; 10-14 Moderate depression; 15-19 Moderately severe depression; 20-27 Severe depression.
Depression Severity | 12 Month Follow Up
  Total scores from the Patient Health Questionnaire (PHQ-9-M) will be used to assess depression severity. Total Score Depression Severity: 0-4 No or Minimal depression; 5-9 Mild depression; 10-14 Moderate depression; 15-19 Moderately severe depression; 20-27 Severe depression.
Suicidal Ideation and Behavior | Baseline
  Suicidal attempt and ideation will be measured through the Columbia Suicide Severity Rating Scale (C-SSRS). The following outcomes are C-SSRS categories: Wish to be Dead; Non-specific Active Suicidal Thoughts; Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Active Suicidal Ideation with Specific Plan and Intent; Preparatory Acts or Behavior; Aborted Attempt; Interrupted Attempt; Actual Attempt (non-fatal); Completed Suicide.
  Self-injurious behavior without suicidal intent is also a C-SSRS outcome and has a binary response (yes/no).
  Suicidal Ideation Score is a numerical score derived from the C-SSRS categories. The maximum suicidal ideation category (1-5 on the CSSRS) present at the assessment. Assign a score of 0 if no ideation is present.
Suicidal Ideation and Behavior | 1 month follow up
  Suicidal attempt and ideation will be measured through the Columbia Suicide Severity Rating Scale (C-SSRS). The following outcomes are C-SSRS categories: Wish to be Dead; Non-specific Active Suicidal Thoughts; Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Active Suicidal Ideation with Specific Plan and Intent; Preparatory Acts or Behavior; Aborted Attempt; Interrupted Attempt; Actual Attempt (non-fatal); Completed Suicide.
  Self-injurious behavior without suicidal intent is also a C-SSRS outcome and has a binary response (yes/no).
  Suicidal Ideation Score is a numerical score derived from the C-SSRS categories. The maximum suicidal ideation category (1-5 on the CSSRS) present at the assessment. Assign a score of 0 if no ideation is present.
Suicidal Ideation and Behavior | 3 month follow up
  Suicidal attempt and ideation will be measured through the Columbia Suicide Severity Rating Scale (C-SSRS). The following outcomes are C-SSRS categories: Wish to be Dead; Non-specific Active Suicidal Thoughts; Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Active Suicidal Ideation with Specific Plan and Intent; Preparatory Acts or Behavior; Aborted Attempt; Interrupted Attempt; Actual Attempt (non-fatal); Completed Suicide.
  Self-injurious behavior without suicidal intent is also a C-SSRS outcome and has a binary response (yes/no).
  Suicidal Ideation Score is a numerical score derived from the C-SSRS categories. The maximum suicidal ideation category (1-5 on the CSSRS) present at the assessment. Assign a score of 0 if no ideation is present.
Suicidal Ideation and Behavior | 6 month follow up
  Suicidal attempt and ideation will be measured through the Columbia Suicide Severity Rating Scale (C-SSRS). The following outcomes are C-SSRS categories: Wish to be Dead; Non-specific Active Suicidal Thoughts; Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Active Suicidal Ideation with Specific Plan and Intent; Preparatory Acts or Behavior; Aborted Attempt; Interrupted Attempt; Actual Attempt (non-fatal); Completed Suicide.
  Self-injurious behavior without suicidal intent is also a C-SSRS outcome and has a binary response (yes/no).
  Suicidal Ideation Score is a numerical score derived from the C-SSRS categories. The maximum suicidal ideation category (1-5 on the CSSRS) present at the assessment. Assign a score of 0 if no ideation is present.
Suicidal Ideation and Behavior | 12 month follow up
  Suicidal attempt and ideation will be measured through the Columbia Suicide Severity Rating Scale (C-SSRS). The following outcomes are C-SSRS categories: Wish to be Dead; Non-specific Active Suicidal Thoughts; Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Active Suicidal Ideation with Specific Plan and Intent; Preparatory Acts or Behavior; Aborted Attempt; Interrupted Attempt; Actual Attempt (non-fatal); Completed Suicide.
  Self-injurious behavior without suicidal intent is also a C-SSRS outcome and has a binary response (yes/no).
  Suicidal Ideation Score is a numerical score derived from the C-SSRS categories. The maximum suicidal ideation category (1-5 on the CSSRS) present at the assessment. Assign a score of 0 if no ideation is present.

SECONDARY OUTCOMES:
Service Utilization | Baseline
  Frequency and type of concurrent psychiatric services will be measured through the Child and Adolescent Services Assessment (CASA).The CASA is a semi-structured face-to-face interview. The interview mixes close-ended questions that are often answered by "yes" or "no" with open-ended questions that allow elaboration. The CASA is comprised of four sections: The Child Health Services Screen, The Detailed Child Services Form, Attitudes Toward Services for Children and Adolescents, and Family Demographic and Financial Information (in the parent version only).
Service Utilization | 6 month follow up
  Frequency and type of concurrent psychiatric services will be measured through the Child and Adolescent Services Assessment (CASA).Frequency and type of concurrent psychiatric services will be measured through the Child and Adolescent Services Assessment (CASA).The CASA is a semi-structured face-to-face interview. The interview mixes close-ended questions that are often answered by "yes" or "no" with open-ended questions that allow elaboration. The CASA is comprised of four sections: The Child Health Services Screen, The Detailed Child Services Form, Attitudes Toward Services for Children and Adolescents, and Family Demographic and Financial Information (in the parent version only).
Service Utilization | 12 month follow up
  Frequency and type of concurrent psychiatric services will be measured through the Child and Adolescent Services Assessment (CASA).Frequency and type of concurrent psychiatric services will be measured through the Child and Adolescent Services Assessment (CASA).The CASA is a semi-structured face-to-face interview. The interview mixes close-ended questions that are often answered by "yes" or "no" with open-ended questions that allow elaboration. The CASA is comprised of four sections: The Child Health Services Screen, The Detailed Child Services Form, Attitudes Toward Services for Children and Adolescents, and Family Demographic and Financial Information (in the parent version only).
Application Utilization | Post-intervention-6 month follow up
  Use of the technical components of interventions and web portals of iCHART including: the number and proportion of adolescents, parents, and providers who have engaged with the application over time
Intervention Acceptability (intervention liked by study population) | Post-intervention-6 month follow up
  Acceptability of the iCHART intervention will be assessed through the 4 item Acceptability of Intervention Measure (AIM). Scales can be created for by averaging responses. Scale values range from 1 to 5. Higher scores indicate greater acceptability. The items include questions to determine if intervention is appealing to, liked by, welcomed by, and approved by study population.
Intervention Usability | Post-intervention-6 month follow up
  Usability of the iCHART intervention will be assessed through the Post System Satisfaction Usability Questionnaire (PSSUQ). PSSUQ follows a 7-point Likert Scale (+ NA option). The overall result is calculated by averaging the scores from the 7 points of the scale. It also has 3 sub-scales, namely system usefulness, information quality, and interface quality. The sub-scales provide a more detailed breakdown of different factors affecting the intervention. PSSUQ score starts with 1 (strongly agree) and ends with 7 (strongly disagree). The lower the score, the better the performance and satisfaction.
Intervention Feasibility (intervention is implementable in study population) | Post-intervention-6 month follow up
  Feasibility of the iCHART intervention will be assessed through the 4 item Feasibility of Intervention Measure (FIM). Scales can be created for by averaging responses. Scale values range from 1 to 5. Higher scores indicate greater feasibility. The items include questions to determine if intervention is easy to use and seems possible or doable to implement in study population.
Intervention Appropriateness (intervention fits or matches study population needs) | Post-intervention-6 month follow up
  Intervention appropriateness of the iCHART intervention will be assessed through 4 item Intervention Appropriateness Measure (IAM). Scales can be created for by averaging responses. Scale values range from 1 to 5. Higher scores indicate greater appropriateness. The items include questions to determine if intervention is a good match, fitting, suitable, or seems applicable to the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Stepp, PhD, Principal Investigator — University of Pittsburgh
Locations (13):
- United States (13):
  - Gibbsboro, Gibbsboro, New Jersey
  - Conemaugh Memorial Medical Center-Family Medicine, Johnstown, Pennsylvania
  - CHOP Primary Care, CHOP Campus, Philadelphia, Pennsylvania
  - Roxborough, Philadelphia, Pennsylvania
  - CHOP Primary Care, Cobbs Creek, Philadelphia, Pennsylvania
  - Karabots, Philadelphia, Pennsylvania
  - Children's Community Pediatrics (CCP) of Children's Hospital of Pittsburgh UPMC, Pittsburgh, Pennsylvania
  - UPMC Center for Adolescent and Young Adult Health, Pittsburgh, Pennsylvania
  - UPMC Family Medicine, Pittsburgh, Pennsylvania
  - Kids Plus Pediatrics (KPP), Pittsburgh, Pennsylvania
  - Berks Community Health Center, Reading, Pennsylvania
  - Springfield, Springfield, Pennsylvania
  - CHOP Primary Care, West Chester, West Chester, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
All requests for study data will follow NIMH's data sharing and data use policies. The final completely de-identified dataset(s) will include demographic and clinical data at baseline, and primary and secondary outcomes for all studies, including those funded by the innovation contests. These analytic datasets may also include derived variables with documentation. Our form datasets will include original case report forms, a detailed codebook of variable names, value labels, and programming formats and all study documentation including the protocol and manual of procedures. For descriptive/raw data, study investigators/study staff will upload to NIMH's National Database for Clinical Trials Related to Mental Health Illness (NDCT) on a semi-annual basis all analyzed data being uploaded prior to primary paper publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following "main outcomes" article publications.
Access Criteria: In addition to public access to the NDCT, proposals should be directed to georgeba2@upmc.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years.

DOCUMENTS (1):
  • Informed Consent Form (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT05748730/ICF_000.pdf